CLINICAL TRIAL: NCT05930743
Title: Climate Change Resilience of Indigenous SocioEcological Systems: RISE
Brief Title: Climate Change Resilience of Indigenous SocioEcological Systems
Status: Completed | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: MU-CIRB2021/227.3004
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Nutrition, Healthy

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The RISE project aims to understand how future climate change may compromise traditional food systems (TFS) by altering related human-nature interactions. A comparative case study approach coupling on-site socioeconomic, nutritional, and ecological surveys of the target indigenous socioecological systems (ISES) of Karen (Kanchanaburi, Thailand) and Sakha (Republic of Sakha, Russian Federation) people with statistical models projecting future changes in the distribution and composition of traditional food species under contrasting climate change scenarios.

DETAILED DESCRIPTION:
The UN Declaration on the Rights of Indigenous Peoples (IPs) recognizes "the right to the lands, territories, and resources which IPs have traditionally owned, occupied or otherwise used or acquired." Within this context, food sovereignty and the sustainability of TFS are emergent issues within the sustainable development agenda as recognized by the United Nations Permanent Forum of Indigenous Peoples' Issues (UNPFII). However, IPs are especially vulnerable to climate change and other environmental impacts. Disrupted ISES are characterized by increased food insecurity and inequalities, loss of traditional identity, westernization of livelihoods, and nutritional problems. The degree of vulnerability to these factors depends upon their adaptation capacity and resilience. Understanding the complex relationships among climate change, socioeconomic development, and TFS is crucial for informing adaptive strategies and promoting the sustainability of ISS in line with international agendas such as the Paris Agreement and the 2030 Sustainable Development Goals (SDGs).

The movement for development emphasizes collaboration among various partners to deal with climate change effectively and to strengthen people's capacity to cope with present and future threats. Thailand has addressed relevant agenda to transform missions in response to climate change as the movement to establish food security based on the sufficient economic principle, the promotion of sustainable agricultural development, the encouragement of good food manufacturing, empowerment of health impact management, and the protection of biodiversity to reenergize natural ecosystem sustainability, for instances.

RISE aims at bridging this gap by using a novel, transdisciplinary risk assessment framework in a comparative case study context using two contrasting ISES: the Karen people, the most indigenous ethnic minority of Thailand, and indigenous communities of the Sakha Republic (Yakutia) in Siberia. The Arctic and Tropics are sentinels and harbingers of climate and environmental change. They are home to a significant proportion of the world's IPs and face some of the most unprecedented, pressing anthropogenic and environmental impacts.

Multiple components of the research study include the following studies. 1) Socioeconomic analysis of indigenous socioecological systems 2) Nutritional/dietary analysis of Indigenous Socioecological Systems 3) Project future changes in traditional food systems from contrasting scenarios of climate change and socioeconomic development 4) Estimate the risk to ISES sustainability and explore limits and enablers of adaptation to inform regional development and the climate and sustainably policy agendas.

ELIGIBILITY:
Inclusion Criteria:

* School-aged children 6-12 years old who are the Karen living in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand
* Working adults 19-59 years old
* who are the Karen living in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand
* with no history of mental illness that has been diagnosed by a doctor, such as schizophrenia, delusional psychosis, bipolar disorder, acute mental illness, psychosis caused by physical disease, and psychosis caused by various substances or drugs.
* who do not have serious underlying diseases such as heart disease, or cancer, which are specified by a doctor and are advised to eat a therapeutic diet.
* Elderly aged 60 and over
* who are the Karen living in Laiwo Subdistrict, Sangkhlaburi District, Kanchanaburi Province, Thailand
* with no history of mental illness that has been diagnosed by a doctor, such as schizophrenia, delusional psychosis, bipolar disorder, acute mental illness, psychosis caused by physical disease, and psychosis caused by various substances or drugs.
* who do not have serious underlying diseases such as heart disease, or cancer, which are specified by a doctor and are advised to eat a therapeutic diet.

Exclusion Criteria:

* Participants who are seriously ill, such as accidents, symptoms from underlying diseases, or other diseases during the data collection are unable to conduct an interview.
* Participants who were out of the village during the data collection period are unable to provide information to the research team.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The indigenous group of Karen people stays in Thungyai - Huai Kha Khaeng Wildlife Sanctuary, the area in the west of Kanchanaburi Province. The population data of the two villages, Saneaphong and Koh Sadueng, were surveyed in 2021. Three aspects of nutritional assessment will compose of three groups of local people according to age range, including (i) school-aged children (6 - 12 y), (ii) adults (19 - 59 y), and (iii) elderly (60 y and over). The population of Saneaphong and Koh Sadueng were 696 and 262 people, respectively. Then the sample size in each village was calculated using the Taro Yamane formula, 1973.
Sampling Method: Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Dietary intake assessment (24-hour dietary recall) | 1 month
  The 24-hour dietary recall interview will be conducted on a single day in both rainy and dry seasons. The resulting data will be analyzed for energy and nutrient intakes using the INMUCAL Nutrients v4 program (INMU, Thailand). Differences in nutritional composition between traditional and market food will be investigated.
Dietary intake assessment (food frequency questionnaire (FFQ)) | 1 month
  A food frequency questionnaire or checklist of specific food items will be developed to determine seasonal food consumption patterns. Data collection will be conducted in both rainy and dry seasons.

SECONDARY OUTCOMES:
Biochemical assessment | 5 days
  Biochemical assessment from venous blood samples taken after a 12-h overnight fast. Blood samples will be transferred to the hospital laboratory for biochemical analysis. Whole blood samples in EDTA vacutainer will be analyzed for complete blood count using automated analyzer. Other blood samples will be centrifuged and analyzed for lipid profile including total cholesterol, high density lipoprotein cholesterol, low density lipoprotein cholesterol and triglycerides using enzymatic colorimetric technique.

OTHER OUTCOMES:
measurement of height | 5 days
  measuring height using a portable stadiometer (unit: centimeter)
measurement of body weight | 5 days
  measuring body weight using a portable bioelectrical impedance scale (unit: kilogram)
measurement of percentage of body fat | 5 days
  measuring the percentage of body fat using a portable bioelectrical impedance scale (unit: percent)
Adult Body Mass Index (BMI) | 5 days
  BMI (unit: kg/m^2) will be calculated from participants' measured weight and height, whereas BMI for age will be considered for children aged 5-19 years according to their nutritional status.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanaephong and Koh Sadueng, Kanchanaburi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sirisai S, Chotiboriboon S, Sapsuwan C, Tantivatanasathien P, Setapun N, Duangnosan P, Thongkam N, Chuangyanyong S. Matriarchy, Buddhism, and food security in Sanephong, Thailand. Matern Child Nutr. 2017 Nov;13 Suppl 3(Suppl 3):e12554. doi: 10.1111/mcn.12554. PMID 29359429
- [Background] Azais-Braesco V, Goffi C, Labouze E. Nutrient profiling: comparison and critical analysis of existing systems. Public Health Nutr. 2006 Aug;9(5):613-22. doi: 10.1079/phn2006966. PMID 16923293
- See also: Indigenous People's Food Systems: the many dimensions of culture, diversity and environment for nutrition and health — https://www.fao.org/documents/card/es/c/250ee74b-9c3f-5dc1-8086-6e0b78b22795